CLINICAL TRIAL: NCT04190290
Title: Efficacy of Adapted Program of Physiotherapy in Hospitalized Person by Anorexia Nervosa With Several Undernutrition
Brief Title: Anorexia Nervosa Inpatient Physiotherapy Adapted Program
Acronym: ANIPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Emilio José Miñano Garrido, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMU
Record Dates: First submitted 2019-11-22; First posted 2019-12-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Muscle strength; Peak-expiratory-flow; Quality of life
MeSH Terms: conditions — Anorexia Nervosa | interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: Quasi experimental prospective study
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mobilizations and exercises training Respiratory exercises Body image exercises
  Interventions: Other: Physiotherapy Adapted Program; Diagnostic Test: Evaluation and Control
- Control (Active Comparator): Muscle strength evaluation and Eating behavior evaluation and Quality of life
  Interventions: Diagnostic Test: Evaluation and Control

INTERVENTIONS:
Other: Physiotherapy Adapted Program — 3 days / week mobilisations and respiratory exercises and body image exercises
  Other Names: Adapted exercises
  Arms: Intervention
Diagnostic Test: Evaluation and Control — Manual muscle test MRC score, peak-expiratory-flow test, hand strength test, 6 minutes walking test, SF-36, EDI-3 and EDQOL

SUMMARY:
Anorexia nervosa (AN) is a psychiatric pathology with several somatics consequences that increase the vital risk. The prevalence in AN is between 0.9-3% and AN has the most elevated mortality in the psychiatric pathologies (10% in the hospitalized patients).

The collateral effects by several undernourishment has been studied but the autonomy and muscle strength research is insufficient.

Physiotherapy research study body image, basic body awareness therapy, relaxation and quality of life.

DETAILED DESCRIPTION:
OBJETIVE: Develop a physiotherapy program to increase muscle strength and quality of life in anorexia nervosa hospitalized patients.

METHOD: 4 weeks of adapted exercises (3 days/week) in anorexia nervosa patients with body max index under 16 in interventional group.

And evaluation program once a week in interventional group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Hospitalized
* Anorexia nervosa
* Body mass index (kg/m2) < 16

Exclusion Criteria:

* Men

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Strength | 4 weeks
  Muscle strength with Manual Muscle Test MRC Scale (0 no articular motion/no muscle contraction. 5 complete articular motion/normal muscle resistance) and hand strength in kilogrammes and Peak Expiratory Flow level in litres/minute
Resistance | 4 weeks
  Cardiopulmonary function with six minute walking test. Calculate the distance walked in 6 minutes in metres.
Life | 4 weeks
  The Short Form Health Survey test (SF-36) is a patient-reported survey of patient health. Spanish version with 36 questions.
  Eating Disorders Quality of Life test (EDQOL) is a simple questionnaire with 25 questions (9 psychological, 6 physical/cognitive, 5 financial, 5 work/school).
Behavior | 4 weeks
  Eating disorders inventory (EDI-3). This test is a self-report questionnaire used to assess the presence of eating disorders. The test has 12 items: 3 items specific of eating disorders (thinness obsession, bulimia, body dissatisfaction) and 9 psychological items (self esteem, personal alignment, interpersonal insecurity, interpersonal distrust, deficit introspective, emotional disturbance, perfectionism, asceticism, fear of maturity)

SECONDARY OUTCOMES:
Others | 4 weeks
  Biological data (potassium, transaminases), weight in kilogrammes and body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Reina Sofía, Murcia, Spain